CLINICAL TRIAL: NCT02486198
Title: Monosialotetrahexosylganglioside Sodium Injection for Treatment of Oxaliplatin Induced Neurotoxicity in Gastrointestinal Cancer
Brief Title: Monosialotetrahexosylganglioside for Treatment of Oxaliplatin Induced Neurotoxicity in Gastrointestinal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TianjinCIH20141201
Record Dates: First submitted 2015-05-03; First posted 2015-07-01 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2015-05

CONDITIONS: Neurotoxicity
Keywords: Gastrointestinal cancer; oxaliplatin; neurotoxicity
MeSH Terms: conditions — Neurotoxicity Syndromes; Gastrointestinal Neoplasms | interventions — Sodium Chloride; Oxaliplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo+oxaliplatin-based chemotherapy (Placebo Comparator): equal saline as placebo, one hour before chemotherapy (if with chemotherapy) with oxaliplatin-based chemotherapy (every 2 or 3 weeks), or daily use until neurotoxicity progress.
  Interventions: Drug: placebo; Drug: oxaliplatin-based chemotherapy
- GM+oxaliplatin-based chemotherapy (Experimental): monosialotetrahexosylganglioside Sodium Injection, 40mg or 60mg, one hour before chemotherapy (if with chemotherapy) with oxaliplatin-based chemotherapy (every 2 or 3 weeks), or daily use until neurotoxicity progress.
  Interventions: Drug: GM; Drug: oxaliplatin-based chemotherapy

INTERVENTIONS:
Drug: placebo — 1. For patients with oxaliplatin-based chemotherapy(every 2 or 3 weeks), equal saline as placebo should be used one hour before oxaliplatin for 1 week during every chemotherapy cycle, until neurotoxicity progressed.
  2. For patients who discontinue oxaliplatin-based chemotherapy, equal saline as placebo should be used daily until there is no neurotoxicity relief (neurotoxicity should be assessed at 2 and 4 weeks' treatment, up to 18 weeks)
  Other Names: Saline
  Arms: placebo+oxaliplatin-based chemotherapy
Drug: GM — 1. For patients with oxaliplatin-based chemotherapy(every 2 or 3 weeks), monosialotetrahexosylganglioside sodium injection(40mg for chemotherapy of every 2 weeks or 60mg for chemotherapy of every 3 weeks)should be used one hour before oxaliplatin for 1 week during every chemotherapy cycle, until neurotoxicity progressed.
  2. For patients who discontinue oxaliplatin-based chemotherapy, equal monosialotetrahexosylganglioside sodium injection should be used daily until there is no neurotoxicity relief (neurotoxicity should be assessed at 2 and 4 weeks' treatment, up to 18 weeks)
  Other Names: Brand name: shenjie
  Arms: GM+oxaliplatin-based chemotherapy
Drug: oxaliplatin-based chemotherapy — chemotherapy contains oxaliplatin
  Other Names: eloxatin,aiheng

SUMMARY:
The purpose of this study is to determine whether Monosialotetrahexosylganglioside sodium injection can relieve the neurotoxicity caused by oxaliplatin in GI cancer.

DETAILED DESCRIPTION:
Oxaliplatin is widely used in GI cancer. Neutropenia and neurotoxicity are the most common adverse effects of oxaliplatin which even result in discontinue of chemotherapy, especially for patients suffered from heavily acute neurotoxicity.The continuous sense and/or motor abnormal reduce the quality of life. To date, there is no a drug to treat oxaliplatin induced neurotoxicity. Monosialotetrahexosylganglioside(GM) is a component of membrane of nerve cells. Previous phase II clinical trial showed, it can reduce oxaliplatin-induced neurotoxicity (OIN). But it did not investigated for curing OIN in randomized control trial. A phase III trial is needed to investigate the effect and safety of monosialotetrahexosylganglioside Sodium Injection for treatment OIN at GI cancer. Investigators design this randomized phase III placebo-controlled trail to identify the effect of monosialotetrahexosylganglioside sodium injection as a treatment agent for OIN. Investigators found 2.5% patients of grade 2 or more serious OIN would relieve with 3 months(data not published). Investigators assume monosialotetrahexosylganglioside can reduce neurotoxicity by 30%. At the level of power 0.8, the sample size is 160 with 10% dropout. If there is no dropout, the trial will be terminated at 144 events occur.The board of Tianjin cancer hospital has permitted the trial and will monitor the whole process of this study. All data will be submitted to the department of clinic trials at Tianjin cancer hospital.The statistics specialist is participating this design and will afford help for data analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients shall have normal organic function such as liver function, Cardiac function and renal function;
2. male or female age >18 years old;
3. diagnosis GI cancer with histology;
4. Chronic neurotoxicity grade is 2 or more
5. Karnofsky Performance scores should be 80 or more
6. patients are in oxaliplatin-based chemotherapy courses or no more than 21 days after last oxaliplatin usage for patients who will discontinue oxaliplatin usage.
7. without uncured tumor except GI cancer,
8. Patients should be expected to live no shorter than 3 months

Exclusion Criteria:

1. patients who is receiving anti-neurotoxicity treatment;
2. WBC<4.0×109/L，ANC<1.5×109/L,PLT<100×109/L，Hb<90g/L,TBIL>1.5Limitation;BUN）>1.5Limitation；Cr）>1.5Limitation；ALT or AST>2.5Limitation（without liver metastasis）；ALT or AST）>5Limitation（with liver metastasis）;
3. heart dysfunction;
4. brain metastasis with symptoms;
5. peripheral nervous system or central nervous system abnormal including diabetes mellitus patients with neuropathy;
6. in situation of oxaliplatin-based chemotherapy progressed, the next chemotherapy regime should not contain agents which will cause neurotoxicity (such as paclitaxel and cisplatin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2015-05-05 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
The relief of neurotoxicity in patients with grade 2 or higher neurotoxicity by means of CTC 4.03 and EORTC QLQ-CIPN20 | From the time recruited to neurotoxicity progressed(assesse before chemotherapy) or without relief(assess at week 2 and 4, up to 18 weeks)
  Besides CTC 4.03 and modified EORTC QLQ-CIPN20, patients will evaluate the neurotoxicity relief extent on the Visual Analog Scale

SECONDARY OUTCOMES:
Safety of Monosialotetrahexosylganglioside sodium injection in treatment of Oxaliplatin induced Neurotoxicity in Gastrointestinal cancer as measured by the number of any adverse effect | every 2 or 3 weeks during GM usage and will continue to assess every 3 months, up to 1 year
  The number of any adverse effect will be used to assess safety
quality of life | evaluate 1 week before interventions'usage and every 4 weeks , up to 24 weeks. And evaluate once within 4 weeks after the patients out of the study
  investigators use sf-36 to evaluated the quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ba, MD.PHD, Principal Investigator — Tianjin Cancer Hospital
Locations (1):
- TianjinCIH, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Zhou L, Liu R, Huang D, Li H, Ning T, Zhang L, Ge S, Bai M, Wang X, Yang Y, Wang X, Chen X, Gao Z, Luo L, Yang Y, Wu X, Deng T, Ba Y. Monosialotetrahexosylganglioside in the treatment of chronic oxaliplatin-induced peripheral neurotoxicity: TJMUCH-GI-001, a randomised controlled trial. EClinicalMedicine. 2021 Oct 29;41:101157. doi: 10.1016/j.eclinm.2021.101157. eCollection 2021 Nov. PMID 34765950